CLINICAL TRIAL: NCT01742455
Title: Quantitative Assessment of the Peripheral Artery Collateral Circulation in Patients With and Without Coronary Artery Disease (Pilot Study)
Brief Title: Assessment of Natural Bypasses in the Lower Limb
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Heart Foundation (Other); Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Christian Seiler, Professor and Co-Chairman of Cardiology, Insel Gruppe AG, University Hospital Bern
Other Study IDs: 256/09
Record Dates: First submitted 2012-11-27; First posted 2012-12-05 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Peripheral Collaterals; Arteriogenesis; Coronary Artery Disease
Keywords: Peripheral artery disease; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Arteriosclerosis; Pathologic Processes
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Myocardial Ischemia; Arteriosclerosis; Pathologic Processes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (routine)
Oversight: Data Monitoring Committee: No

SUMMARY:
Concerning the promotion of peripheral collateral growth, clinical studies investigating new therapeutic strategies have used imprecise assessment methods and therefore determined only "weak" endpoints. In contrast to the coronary circulation, there is currently no gold standard available to document successful promotion of collateral growth in patients suffering from peripheral artery disease. Therefore, the purpose of this study is to evaluate a new invasive method to quantify arterial collateral flow in the lower extremity in patients undergoing elective coronary angiography.

DETAILED DESCRIPTION:
Background: Peripheral artery disease (PAD) of the lower extremities is due to arterial obstruction leading to reduced arterial flow during exercise and/or at rest. The disease is present in approximately 4 percent of persons >40 years of age, but in 15-20 percent of those >65 years. Claudication is the major symptom and can improve with pharmacotherapy or exercise rehabilitation. In patients with disabling claudication that persist despite exercise and pharmacotherapy or with critical limb ischemia (i.e. ischemic rest pain; ulcers or gangrene at risk of major amputation), revascularization therapies are indicated. However, in about 1/4 of these patients endovascular or surgical therapy fails or is not applicable, making alternative approaches necessary.1 Thus, promotion of angiogenesis, a process triggered by ischemia with sprouting of capillaries insufficient to provide adequate blood supply to jeopardized tissues, and arteriogenesis, which refers to positive remodeling of preformed collateral arterioles, i.e. collateral growth should be applied in these patients.2, 3 Despite the fact that numerous studies during the last decade pursued the important therapeutic strategy of improving collateral function in patients with PAD, there is currently no method available to quantify collateral arterial function of the lower limb and, thus, to determine therapeutic effects. Clinical studies investigating new therapeutic strategies for the promotion of peripheral collateral growth by application of growth factors and/or exercise rehabilitation have used imprecise and inadequate assessment methods and therefore determined only "weak" endpoints. In contrast to the coronary circulation, there is currently no gold standard available to document successful promotion of collateral growth in patients suffering from PAD.

Aim: The purpose of this study in patients undergoing elective coronary angiography with or without chronic stable coronary artery disease is to evaluate a new invasive method to quantify arterial collateral flow in the lower extremity.

Main hypothesis: Quantitative assessment of peripheral arterial collaterals by pressure-derived collateral flow index (CFIp) in the lower extremities is safe and feasible.

Methodology: Prospective exploratory trial. Primary study endpoint: Pressure-derived collateral flow index (CFIp) of the superficial femoral artery.

Potential significance: The results of this study will demonstrate that the concept of collateral flow index - which has been proven by our group in the coronary circulation - is a safe and feasible method for the quantitative assessment of peripheral limb collateral function. The results of this study may serve as preliminary data for larger clinical trials investigating therapeutic promotion of collaterals in patients with PAD and provide a reliable study endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Stable angina pectoris, electively referred for coronary angiography
* Written informed consent to participate in the study

Exclusion Criteria:

* Rest pain, ulceration or gangrene due to PAD (Rutherford 4-6)
* Significant stenoses (>50%) or occlusion of superficial femoral or profunda femoral artery
* Aortoiliac occlusion or significant stenoses (>50%)
* Aneurysm of abdominal aorta or iliac arteries
* Acute coronary syndrome
* Congestive heart failure NYHA III-IV
* Severe pulmonary arterial hypertension
* Severe hepatic or renal failure (creatinine clearance < 15ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients with stable angina pectoris electively referred for coronary angiography to our department who give written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pressure-derived collateral flow index (CFIp) of the superficial femoral artery | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Prof., Study Chair — Insel Gruppe AG, University Hospital Bern; Tobias Traupe, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Seiler C. Collateral Circulation of the Heart. 1st ed. London: Springer-Verlag; 2009.
- [Background] Kalka C, Baumgartner I. Gene and stem cell therapy in peripheral arterial occlusive disease. Vasc Med. 2008;13(2):157-72. doi: 10.1177/1358863x08088616. PMID 18593804
- [Background] De Vivo S, Palmer-Kazen U, Kalin B, Wahlberg E. Risk factors for poor collateral development in claudication. Vasc Endovascular Surg. 2005 Nov-Dec;39(6):519-24. doi: 10.1177/153857440503900609. PMID 16382273
- [Background] van Royen N, Schirmer SH, Atasever B, Behrens CY, Ubbink D, Buschmann EE, Voskuil M, Bot P, Hoefer I, Schlingemann RO, Biemond BJ, Tijssen JG, Bode C, Schaper W, Oskam J, Legemate DA, Piek JJ, Buschmann I. START Trial: a pilot study on STimulation of ARTeriogenesis using subcutaneous application of granulocyte-macrophage colony-stimulating factor as a new treatment for peripheral vascular disease. Circulation. 2005 Aug 16;112(7):1040-6. doi: 10.1161/CIRCULATIONAHA.104.529552. Epub 2005 Aug 8. PMID 16087795
- [Background] Traupe T, Gloekler S, de Marchi SF, Werner GS, Seiler C. Assessment of the human coronary collateral circulation. Circulation. 2010 Sep 21;122(12):1210-20. doi: 10.1161/CIRCULATIONAHA.109.930651. No abstract available. PMID 20855668
- [Derived] Traupe T, Ortmann J, Stoller M, Baumgartner I, de Marchi SF, Seiler C. Direct quantitative assessment of the peripheral artery collateral circulation in patients undergoing angiography. Circulation. 2013 Aug 13;128(7):737-44. doi: 10.1161/CIRCULATIONAHA.112.000516. Epub 2013 Jul 1. PMID 23817577